CLINICAL TRIAL: NCT03466853
Title: Assessment by the CANS Score Versus Anthropometry and Impact on Early Neonatal Morbidities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Other Study IDs: 33
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Fetal Malnutrition
MeSH Terms: conditions — Fetal Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Clinical assessment of nutritional status (CANS) score — Systematized inspection and estimation of loss of SC tissues and muscles of nine superficial physical parameters including hair and buccal fat in the cheeks, chin and neck, arms, back, inter or subscapular skin, buttocks, legs, chest, and abdominal wall skin. These signs will be rated from 1 (worst, severe FM) to 4 (best, well nourished), and the highest and lowest total scores are 36 and 9, 3respectively. A total score of <25 is considered as fetal malnutrition.
Diagnostic Test: Anthropometric indices — weight, length and head circumference
Diagnostic Test: Proportionality indices — MAC/HC ratio (Calculation for each infant and value will be plotted on and compared with a standard curve). Ponderal index . A PI <2.2 is considered as malnutrition). Body mass index (BMI= weight (kg) / length2 (m). A BMI <11.2 kg/m2 is considered as malnutrition)

SUMMARY:
Assessment of malnutrition within 48 hours of birth through anthropometric indices as Weight, Length and Head circumference, Proportionality indices as MAC/HC ratio, Ponderal index and Body mass index, Clinical assessment of nutritional status (CANS) score. Detection of early neonatal morbidities within the first week of life including Hypoglycemia ,Polycythemia, Respiratory Distress Syndrome, Neonatal sepsis, Hyperbilirubinemia and Feeding intolerance

DETAILED DESCRIPTION:
Within the 1st 48 hours of birth, all live born, singleton neonates with gestational ages between 28-40 weeks will be included in the study after obtaining an informed consent from their legal guardians.

Assessment of malnutrition within 48 hours of birth:

1. Anthropometric indices:

   Weight (using the infant weighing scale). Length (using the infant measuring board). Head circumference (using non-metallic non-stretchable tape).
2. Proportionality indices:

   MAC/HC ratio (Calculation for each infant and value will be plotted on and compared with a standard curve). Ponderal index Body mass index
3. Clinical assessment of nutritional status (CANS) score:

A total score <25 is considered as fetal malnutrition. 3. Detection of early neonatal morbidities within the first week of life (for those who will require NICU admission):

1. Hypoglycemia (Random blood sugar)
2. Polycythemia (Hematocrit level)
3. Respiratory Distress Syndrome
4. Neonatal sepsis (Clinically, Laboratory: CBC with diff., CRP, C/S)
5. Hyperbilirubinemia (Serum bilirubin level, Need of phototherapy or exchange transfusion)
6. Feeding intolerance (Abdominal distension with prominent intestinal loops, Gastric residue more than 3ml/kg before feeding at least 2 times/ day)

ELIGIBILITY:
Inclusion Criteria:

Neonates of both genders. Gestational age between 28-40 weeks. Singleton pregnancies.

Exclusion Criteria:

Presence of congenital anomalies. Infants of diabetic mothers

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All neonates delivered at Kasr Al-Ainy Gynecology and Obstetrics department, Faculty of Medicine, Cairo University within the proposed study duration Within the 1st 48 hours of birth, all live born, singleton neonates with gestational ages between 28-40 weeks will be included in the study after obtaining an informed consent from their legal guardians
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-01-03 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
infant nutritional status | Within the 1st 48 hours of birth
  To compare the assessment of infant nutritional status using the CANS score against anthropometric and proportionality indices

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided